CLINICAL TRIAL: NCT04818151
Title: Anticoagulation Strategies for the Treatment of Acute Venous Thromboembolism in Medicare Fee For-Service Patients With End-Stage Renal Disease Using USRDS Data
Brief Title: Anticoagulation Strategies for Acute Venous Thromboembolism in Patients With End-Stage Renal Disease Using USRDS Data
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00272929; CV185-804 (Other Grant/Funding Number: Bristol Myers Squibb)
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Venous Thromboembolic Disease; Kidney Failure, Chronic
Keywords: Anticoagulation; Apixaban; Warfarin; Heparin; Bleeding; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Hemorrhage | interventions — Warfarin; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- ESRD patients with VTE treated with warfarin: Warfarin as primary treatment of VTE
  Interventions: Drug: Warfarin
- ESRD patients with VTE treated with apixaban: Apixaban as primary treatment of VTE
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Warfarin — Warfarin treatment for VTE
  Groups: ESRD patients with VTE treated with warfarin
Drug: Apixaban — Apixaban treatment for VTE
  Groups: ESRD patients with VTE treated with apixaban

SUMMARY:
Patients with end stage renal disease (ESRD) are at significantly increased risk of thrombosis and bleeding relative to those with normal renal function which makes anticoagulation particularly challenging. Further, ESRD patients undergoing initiation of anticoagulation for acute VTE are often kept in the hospital for heparin "bridging" which may lead to a protracted length-of-stay (LOS) and may place patients at risk for hospital-associated complications. The advent of direct oral anticoagulants (DOACs) has offered physicians choices in the management of venous thromboembolism (VTE). However, evidence suggests that rivaroxaban and dabigatran are associated with a higher risk of bleeding in ESRD patients. In contrast, research suggests that apixaban may be safer in patients with ESRD, and recent evidence suggests lower bleeding rates in ESRD patients treated for atrial fibrillation with apixaban compared to those treated with warfarin. However, to date, no large national cohort studies have examined the safety, effectiveness, and healthcare utilization of apixaban in patients with ESRD who have acute VTE. The investigators propose to use the Standard Analytic Files from the United States Renal Data System (USRDS) for years 2014 through 2018 to evaluate the safety, effectiveness, and healthcare utilization of ESRD patients initiated on apixaban compared to those initiated on warfarin (following heparin) to treat acute VTE.

DETAILED DESCRIPTION:
The investigators will perform a retrospective cohort analysis using USRDS data from 2014 through 2018 and a descriptive serial cross-sectional analysis using USRDS data from 2009 through 2018 to evaluate the investigators' aims. USRDS data will be utilized to address all the research aims.

Primary Objective To compare rates of major bleeding attributable to initiation of treatment with apixaban relative to warfarin among patients with ESRD and acute VTE The primary safety outcome will be rates of major bleeding within 6 months of VTE diagnosis as defined by Cunningham, which is a standardized definition of major bleeding that can be derived from administrative data and is based on clinical bleeding definitions from a number of clinical trials. A secondary safety outcome will be gastrointestinal bleeding within 6 months of VTE diagnosis.

Secondary Objectives To describe contemporary anticoagulation strategies to treat acute VTE in ESRD patients and changes over the last decade The investigators will report rates of use of anticoagulation strategies [warfarin, low molecular weight heparin (LMWH), and DOACs (apixaban, edoxaban, rivaroxaban, and dabigatran)] in this ESRD population. The investigators will examine rates of these strategies by year to examine changes in adoption of various strategies over time as DOACs have become available for VTE treatment.

To compare rates of recurrent VTE attributable to initiation of treatment with apixaban relative to warfarin among patients with ESRD and acute VTE The primary outcome will be recurrent VTE within 6 months of VTE diagnosis. All-cause mortality within 6 months of VTE diagnosis will be evaluated as an exploratory endpoint.

To compare healthcare resource utilization from 15 days before to 90 days after first prescription date attributable to initiation of treatment with apixaban relative to warfarin among patients with ESRD and acute VTE The primary outcome will be total inpatient days from 15 days before to 90 days after first prescription date. In addition to total inpatient days, the investigators will also compare emergency department (ED) utilization after initiation of anticoagulation across treatment strategies. By incorporating 15 days prior to first prescription date, the investigators will capture hospitalization days that were associated with the index VTE diagnosis, given that the first anticoagulation prescription would likely be written at the time of hospital discharge for those patients who are hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* ESRD on dialysis with acute VTE

Exclusion Criteria:

* Anticoagulation for non-VTE indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in USRDS dataset from 2009-2018 with ESRD and VTE
Sampling Method: Non-Probability Sample
Enrollment: 14914 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Bleeding occurrence | 3 months
  Number of bleeding occurrences.
Recurrent thrombosis occurrence | 3 months
  Number of recurrent thrombosis occurrences.

SECONDARY OUTCOMES:
Days in acute care | 3 months
  Number of hospital days/ED utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Brotman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided